CLINICAL TRIAL: NCT01479660
Title: Probiotic for the Restoration of Intestinal Permeability and Reduction of Intestinal Inflammation in Active Ulcerative Colitis: A Double Blind Randomized Placebo Controlled Trial
Brief Title: Role of Healthy Bacteria in Ulcerative Colitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Collaborators: Ministry of Science and Technology, India (Other Government)
Responsible Party: Principal Investigator, Dr. Bikash Medhi, MBBS, MD(AIIMS),MAMS,FIMSA, Additional Professor, Department of Pharmacology, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11/6095 dated 15/03/2011; CTRI/2011/08/001944 (Registry Identifier: Clinical Trials Registry- India)
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2011-11-24 (Estimated); Status verified 2011-11

CONDITIONS: Ulcerative Colitis
Keywords: Probiotics; ulcerative colitis; inflammatory bowel disease
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator)
  Interventions: Other: Control
- Probiotic (Experimental)
  Interventions: Drug: Probiotic

INTERVENTIONS:
Other: Control — Placebo will be orally administered daily for a period of 12 weeks in high dose and low dose
  Arms: Control
Drug: Probiotic — Probiotic Capsules (450 billion CFU) will be orally administered daily for a period of 12 weeks and Probiotic in higher dose of (3600 billion CFU) will be administered daily for a period of 12 weeks
  Arms: Probiotic

SUMMARY:
Intestinal inflammation seen in inflammatory bowel disease (IBD) results from an altered mucosal immune response to luminal bacterial antigens. Current research suggests that an inappropriate and persistent immune response against commensal intestinal bacterial flora plays a pivotal role in the pathogenesis of chronic Inflammatory Bowel Disease (IBD). It has been also proposed that the signs and symptoms of IBD may be mediated by the increased intestinal permeability secondary to low grade inflammation in the gut mucosa. Increased intestinal permeability results in further exposure of underlying intestinal mucosa to luminal bacteria and antigens perpetuating the intestinal inflammation. Thus restoring intestinal permeability rather than only reduction of mucosal inflammation would thus be a desirable endpoint in the restoration of mucosal integrity and would be the harbinger of better long term outcome. Many clinical trials have shown that probiotics may have beneficial effect on IBD patients. Probiotics are hypothesized to work by several mechanisms though they are not clearly established. The role of probiotics in improving intestinal permeability has not been evaluated. The probiotic VSL #3 is easily available, cheap, effective and safe alternative or substitute for the existing therapeutic agents will be evaluated in this study for their efficacy, tolerability, compliance in inducing clinical response in patients with Ulcerative colitis. This will be a double blind randomized placebo controlled study to determine the clinical efficacy of 12 weeks of oral probiotics (VSL#3) in patients with inflammatory bowel disease. The objectives of this study are to determine the efficacy of probiotics on clinical endoscopic and histological improvement, to find the improvement in faecal, serum and intestinal tissue inflammatory markers, improvement in intestinal permeability, improvement in Quality of life parameters.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Active disease at presentation

Exclusion Criteria:

* Pregnant or lactating women
* Any patient who has received probiotic in the preceding 4 weeks
* Patient with life threatening cardiac, renal, pulmonary or cardiovascular disease
* Inability to obtain the informed consent
* Severe disease requiring hospitalization / steroids/ anti-cytokine therapy
* Patient taking aspirin and other antiplatelet drugs
* Patient with uncontrolled diabetes
* Patient with Gall stone disease
* Patient currently on antibiotic,NSAIDs or indigenous medicine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-10 (Estimated); Study Completion 2014-10 (Estimated)

PRIMARY OUTCOMES:
Reduction of at least 3 points in the D.A.I i.e. Reduction in the activity score of inflammation from the baseline value at 12 weeks. | 12 weeks

SECONDARY OUTCOMES:
Reduction in intestinal permeability | 12 weeks
Reduction in faecal and serum inflammatory markers | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bikash Medhi, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh, India